CLINICAL TRIAL: NCT01506479
Title: Exploratory Study of Different Doses of Endurance Exercise in People With Parkinson Disease
Brief Title: Study in Parkinson's Disease of Exercise
Acronym: SPARX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Illinois at Chicago (Other); University of Pittsburgh (Other); Rush University Medical Center (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-1237; R01NS074343 (NIH)
Record Dates: First submitted 2011-12-16; First posted 2012-01-10 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Basal Ganglia Disease; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases; Brain Diseases
MeSH Terms: conditions — Parkinson Disease; Basal Ganglia Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases; Brain Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (Sham Comparator): Wait listed to moderate or vigorous exercise after 6 months of no exercise.
  Interventions: Behavioral: No Intervention
- Vigorous Exercise (Experimental): Endurance exercise at 80-85% HR max, 4x/wk for 6 months.
  Interventions: Behavioral: Vigorous Exercise
- Moderate Exercise (Experimental): Endurance exercise at 60-65% HR max, 4x/wk for 6 months.
  Interventions: Behavioral: Moderate Exercise

INTERVENTIONS:
Behavioral: Moderate Exercise — Endurance exercise at 60 - 65% heart rate (HR) max,4x/wk for 6 months.
  Arms: Moderate Exercise
Behavioral: Vigorous Exercise — Endurance exercise at 80-85% HR max, 4x/wk for 6 months.
  Arms: Vigorous Exercise
Behavioral: No Intervention — No-exercise control (i.e., usual care);
  Arms: Control Group

SUMMARY:
The purpose of this study is to learn more about the effects of exercise on patients who have been recently diagnosed with Parkinson's disease (PD). The investigators are going to test two levels of exercise (moderate to vigorous) against no exercise. The investigators think that exercise may reduce the symptoms the of PD, and the investigators hope to learn what level of exercise will offer the most benefit.

DETAILED DESCRIPTION:
The overall objective of this study is to determine the futility or non-futility of conducting a randomized controlled trial to determine the effects of exercise on the progression of PD symptoms. The primary aim is to determine whether individuals with de novo Parkinson's disease (naïve to drug treatment) can achieve the randomly assigned levels of mean exercise intensity (60-65% HRmax or 80-85% HRmax) and adhere to the exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary Parkinson's disease
* In a Hoehn and Yahr stage less than stage III
* Disease duration is less than 5 years
* Not likely to require dopaminergic therapy within 6 months

Exclusion Criteria:

* Use of any PD medication within 60 days prior to the beginning the study, including levodopa, direct dopamine agonists, amantadine, Rasagiline (Azilect), Selegiline (Eldepryl), Artane (trihexyphenidyl).
* Duration of previous use of medications for PD that exceeds 90 days
* Expected to require dopaminergic therapy in the next 6 months
* Poorly controlled or unstable cardiovascular disease
* Uncontrolled hypertension
* Hypo- or hyperthyroidism, abnormal liver function, abnormal renal function
* Mild cognitive impairment (Montreal Cognitive Assessment score<26/30)
* Depression that precludes ability to exercise (Beck depression score>13)
* Disorders that interfere with ability to perform endurance exercises
* Regular participation in vigorous endurance exercise
* Evidence of serious arrhythmias or ischemic heart disease
* Any clinically significant medical condition, psychiatric condition, drug or alcohol abuse, or laboratory abnormality that would, in the judgment of the investigators, interfere with the ability to participate in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Schenkman, PT, PhD, Principal Investigator — University of Colorado, Denver; Daniel Corcos, PhD, Principal Investigator — University of Illinois at Chicago
Locations (3):
- United States (3):
  - University of Colorado Denver, Aurora, Colorado
  - University of Illinois, Chicago, Chicago, Illinois
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Hall DA, Moore C, Comella C; SPARX Study Group. Recruitment of patients with de novo Parkinson disease: successful strategies in a randomized exercise clinical trial. Trials. 2018 Nov 14;19(1):630. doi: 10.1186/s13063-018-2958-z. PMID 30428907
- [Derived] Schenkman M, Moore CG, Kohrt WM, Hall DA, Delitto A, Comella CL, Josbeno DA, Christiansen CL, Berman BD, Kluger BM, Melanson EL, Jain S, Robichaud JA, Poon C, Corcos DM. Effect of High-Intensity Treadmill Exercise on Motor Symptoms in Patients With De Novo Parkinson Disease: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):219-226. doi: 10.1001/jamaneurol.2017.3517. PMID 29228079
- [Derived] Moore CG, Schenkman M, Kohrt WM, Delitto A, Hall DA, Corcos D. Study in Parkinson disease of exercise (SPARX): translating high-intensity exercise from animals to humans. Contemp Clin Trials. 2013 Sep;36(1):90-8. doi: 10.1016/j.cct.2013.06.002. Epub 2013 Jun 14. PMID 23770108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prescreening by telephone and for patients in movement disorder clinics from May 2012 to November 2015.
Pre-assignment Details: Screening included confirmation of Parkinson disease diagnosis, assessment of depression and cognition, testing for laboratory measures, and testing for blood pressure and echocardiogram responses to exercise during graded exercise. Once deemed eligible, baseline assessments were completed for disease and non-disease specific scales.
Period: Overall Study
Arm/Group | Control Group | Vigorous Exercise | Moderate Exercise
Started | 40 | 43 | 45
Completed (Number of participants with 6 month follow-up.) | 37 | 38 | 42
Not Completed | 3 | 5 | 3
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Missing assessment | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Vigorous Exercise | Moderate Exercise | Total
Number analyzed (Participants) | 40 | 43 | 45 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10) | 64 (9) | 63 (10) | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 18 | 55
  Male | 24 | 22 | 27 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 6
  Not Hispanic or Latino | 39 | 39 | 41 | 119
  Unknown or Not Reported | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 36 | 39 | 40 | 115
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Unified Parkinson Disease Rating Scale Part 3 Motor Evaluation [Mean (Standard Deviation); unit: units on a scale] — Sum of 27 items scored 0 to 4, minimum score is 0, maximum score is 108. Higher score indicates worse motor symptoms.
  units on a scale | 17 (7) | 17 (7) | 16 (7) | 17 (7)
Total daily steps [Mean (Standard Deviation); unit: steps per day] — Population: Several participants did not wear the activity monitor devices for recording total number of daily steps.
  steps per day
    number analyzed (Participants) | 36 | 36 | 42 | 114
    (all) | 5005 (2987) | 5146 (3107) | 5702 (2521) | 5306 (2856)
Hoehn and Yahr Stage [Count of Participants; unit: Participants] — Stage 1 is Unilateral Disease; Stage 2 is Bilateral Disease without impairment of balance
  Participants
    Stage 1 | 8 | 12 | 13 | 33
    Stage 2 | 32 | 31 | 32 | 95

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Average Maximum Heart Rate During Exercise as a Measure of Adherence to Exercise
Description: To test whether individuals with de novo Parkinson's disease (naïve to drug treatment) can achieve the randomly assigned levels of mean exercise intensity (60-65% average HRmax or 80-85% average HRmax) and adhere to the exercise protocol.
Time Frame: 9 to 26 weeks
Population: Only for participants who contributed heart rate monitor data.
Measure: Mean (95% Confidence Interval); unit: percentage of maximum heart rate
Arm/Group | Vigorous Exercise | Moderate Exercise
Number analyzed (Participants) | 38 | 42
percentage of maximum heart rate | 80.3 [78.8 to 81.7] | 65.9 [64.2 to 67.7]
Statistical Analysis 1: Comparison: Vigorous Exercise vs Moderate Exercise; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 14.3, 95% CI 2-sided [12.0 to 16.6]

2. Secondary Outcome: 6 Month Change in Unified Parkinson's Disease Rating Scale (UPDRS) Motor Score
Description: Participants were assessed at baseline and at 6 months on their UPDRS. If a participant initiated Parkinson disease medication prior to the 6 month assessment, the UPDRS score from the clinical visit assessment prior to this initiation was used as the score for the individual at 6 months. The change in the UPDRS motor score at 6 months was used as the measure for the futility component of the trial. The change at 6 months was measured as the 6 month value minus the baseline score. A positive change represents worsening of motor symptoms; 0 represents no change; negative values represent improvement. The minimum score on the UPDRS motor is 0 and the maximum is 108 at baseline and 6 months with higher scores representing worse motor symptoms.
Time Frame: Baseline and 6 months
Population: Intention to treat; participants were analyzed in the group to which they were assigned. If a participant started medication, the UPDRS measure prior to initiating medication was used even if the 6 month data were not collected. Participants who did not start medications and were missing the 6 month assessment were not included.
Measure: Mean (95% Confidence Interval); unit: units on the UPDRS Motor scale
Arm/Group | Control Group | Vigorous Exercise | Moderate Exercise
Number analyzed (Participants) | 38 | 39 | 42
units on the UPDRS Motor scale | 3.2 [1.4 to 5.1] | 0.3 [-1.7 to 2.3] | 2.0 [0.4 to 3.7]
Statistical Analysis 1: Comparison: Control Group vs Vigorous Exercise; The null hypothesis is that the vigorous exercise group warrants further investigation using a futility threshold of 3.5 compared to the control group (difference between the mean change in the control group and the mean change in the vigorous exercise group). The alternative hypothesis is that vigorous exercise does not warrant further investigation; Test type: Other; p = 0.34, t-test, 1 sided — The a priori threshold for statistical significance was 0.10; Mean Difference (Final Values) = 2.9, 90% CI 1-sided [upper limit 4.6]
Statistical Analysis 2: Comparison: Control Group vs Moderate Exercise; The null hypothesis is that the moderate exercise group warrants further investigation using a futility threshold of 3.5 compared to the control group (difference in the mean change between the control group and the moderate exercise group). The alternative hypothesis is that moderate exercise does not warrant further investigation; Test type: Other; p = 0.03, t-test, 1 sided — The a priori threshold for statistical significance was set to 0.10. If the p-value is less than 0.10, the null hypothesis is rejected in favor of the alternative (moderate exercise does not warrant further investigation); Mean Difference (Final Values) = 1.2, 90% CI 1-sided [upper limit 2.8] — The estimate is the difference between the control group and the moderate exercise group. The upper bound of the confidence interval should be compared to the futility threshold of 3.5 to reject or not reject the null hypothesis

3. Other Pre Specified Outcome: Number of Days of Exercise Per Week
Description: The number of days the participant exercised per week
Time Frame: 9 to 26 weeks
Population: Participants were analyzed in the group to which they were assigned. Participants were not included if they did not start the intervention.
Measure: Mean (95% Confidence Interval); unit: Number of days per week
Arm/Group | Vigorous Exercise | Moderate Exercise
Number analyzed (Participants) | 40 | 45
Number of days per week | 2.8 [2.4 to 3.2] | 3.2 [2.8 to 3.6]
Statistical Analysis 1: Comparison: Vigorous Exercise vs Moderate Exercise; Test type: Superiority; p = 0.1334, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected monthly until the primary time point at 6 months.
Arm/Group | Control Group | Vigorous Exercise | Moderate Exercise
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43 | 2/45
Other Adverse Events (participants affected / at risk) | 13/40 | 28/43 | 24/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=40) | Vigorous Exercise (N=43) | Moderate Exercise (N=45)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=40) | Vigorous Exercise (N=43) | Moderate Exercise (N=45)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 2 (2) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 3 (3)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 9 (11) | 6 (13) | 5 (7)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (9) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No